CLINICAL TRIAL: NCT00263874
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of UK-500,001 Dry Powder For Inhalation (DPI) In Adults With Moderate To Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Phase 2 Study of the Safety and Efficacy of UK-500,001 in Adult Patients With COPD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to terminate was completely related to efficacy and there were no safety concerns.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5641009
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: UK-500,001

SUMMARY:
This initial proof of concept, phase II study aims to assess the safety and efficacy of UK-500,001 for the chronic maintenance treatment of adults with Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-severe COPD (Global inititiative for chronic Obstructive Lung Disease, GOLD, 2003 definition)
* Smoking history of at least 10 pack-years

Exclusion Criteria:

* Any significant co-morbid disease
* Use of any maintenance therapy except short acting bronchodilators

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324
Dates: Start 2005-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Change from baseline in forced expiratory volume in 1 second (FEV1) compared to placebo

SECONDARY OUTCOMES:
Change from baseline in other lung function parameters, dyspnea, quality of life compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Argentina (4):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Vicente López, Buenos Aires
  - Pfizer Investigational Site, Rosario, Santa FÃ©
  - Pfizer Investigational Site, Buenos Aires
- Australia (3):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Canada (4):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Kingston, Ontario
- Chile (3):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago Metropolitan
  - Pfizer Investigational Site, ValparaÃ-so, ValparaÃ-so
- Pfizer Investigational Site, Zagreb, Croatia
- Czechia (4):
  - Pfizer Investigational Site, Olomouc
  - Pfizer Investigational Site, Ostrava-Poruba
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Tábor
- Hungary (3):
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Törökbálint
  - Pfizer Investigational Site, Veszprém
- Pfizer Investigational Site, Singapore, Singapore
- Pfizer Investigational Site, Madrid, Madrid, Spain
- Pfizer Investigational Site, Manchester, United Kingdom

REFERENCES:
- [Derived] Vestbo J, Tan L, Atkinson G, Ward J; UK-500,001 Global Study Team. A controlled trial of 6-weeks' treatment with a novel inhaled phosphodiesterase type-4 inhibitor in COPD. Eur Respir J. 2009 May;33(5):1039-44. doi: 10.1183/09031936.00068908. Epub 2009 Feb 12. PMID 19213793
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5641009&StudyName=Phase+2+Study+of+the+Safety+and+Efficacy+of+UK%2D500%2C001+in+Adult+Patients+with+COPD